CLINICAL TRIAL: NCT05051969
Title: Mindfulness-Based Stress Reduction for Metro Nashville Public School Employees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Martha E. Shepherd, Assistant Professor of Clinical Medicine and Pediatrics, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 211257
Record Dates: First submitted 2021-09-12; First posted 2021-09-21 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Self-compassion; Burnout; Stress; Anxiety; Depression
Keywords: Burnout; Self-compassion
MeSH Terms: conditions — Burnout, Psychological; Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8 Week Remote Mindfulness-Based Stress Reduction Program (Experimental): 8 Week Remote MBSR Course for MNPS Employees.
  Interventions: Behavioral: Remote Mindfulness-Based Stress Reduction Program
- 8 week waitlist control (No Intervention): 8 week waitlist control. They will complete the same assessments at baseline, 8 and 12 weeks

INTERVENTIONS:
Behavioral: Remote Mindfulness-Based Stress Reduction Program — Enrolled participants will participate in a remote-delivered (online with audio and video) Mindfulness-Based Stress Reduction (MBSR) program. MBSR is a well established behavioral health intervention consisting of 10-sessions lasting 2.5 hours, with one session lasting 7.5 hours in an all-day retreat format over a 2-month period.
  Arms: 8 Week Remote Mindfulness-Based Stress Reduction Program

SUMMARY:
Stress, anxiety, and depression are common symptoms among public school teachers. Public school teachers are among the top professions reporting stress, anxiety, and depression. The causes are multifactorial and include work-related demands, challenges with students, limited resources, and compassion fatigue. Because of this, teachers are at risk of burnout and leaving or changing their profession. The COVID-19 pandemic has had a considerable impact on teachers due to disruptions in usual education delivery and ability to support students. Recent reports show poorer mental health and decreases in physical activity in teachers since the onset of the pandemic. Effective and implementable strategies are urgently needed to address poor mental health and to foster positive health characteristics in this population.

Mindfulness programs decrease feelings of stress, anxiety, and emotional exhaustion. Additionally, mindfulness can improve self-compassion, which may be an important mediating factor in a teacher population. Prior work has shown an inverse relationship between self-compassion and burnout. Currently, there are few studies investigating whether building self-compassion can reduce burnout in public school teachers. The investigators will explore therelationship between participation in a Mindfulness-Based Stress Reduction (MBSR) course and changes in burnout, self-compassion, and other whole person health measures in an educator population. The overall objective of this open pilot study is to examine the feasibility and acceptability of an 8-week remote, group-based MBSR program delivered over Zoom for Metro Nashville Public Schools (MNPS) personnel reporting elevated stress, anxiety, and/or depressive symptoms. Our pilot study results will contribute to the evidence on MBSR in a public-school employee population and inform strategies to optimize implementation of our remote MBSR program within the Vanderbilt Health at MNPS system.

ELIGIBILITY:
Inclusion Criteria:

* Working certificated Metro Nashville Public Schools (MNPS) employees who self-report stress, anxiety, and/or depressive symptoms

Exclusion Criteria:

* Unable to commit to the weekly MBSR schedule
* Have taken the MBSR course previously
* Participants who do not have reliable home internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Feasibility - Recruitment | Baseline
  Feasibility of recruitment will be assessed as the number of inviduals who are screened, eligible and enrolled in the study.
Feasibility- class attendance | Baseline to program completion (8 weeks)
  Percentage of participants that attend each scheduled session and who complete the program.
Feasibility- enrollment retention | Baseline to 12 weeks after enrollment
  Retention will be the number and proportion of indviduals who complete patient reported outcome data collection at 12-weeks.
Acceptability - Overall Helpfulness of the course | Baseline to 8 weeks
  Helpfulness of the course assessed by a one question survey with an 11-point Numeric Rating Scale ranging from 0 ("Not helpful") to 10 ("Most helpful"). Lower scores indicate less helpfulness.

SECONDARY OUTCOMES:
Perceived stress as measured by a Perceived Stress Scale | Baseline, 8 weeks and 12 weeks
  10-item Perceived Stress Scale. Each question is scored ranging from 0 (Never) to 4 (Very Often) Total survey scores range from 0-40. A lower score indicates low stress, a better outcome.
Anxiety as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety short form | Baseline, 8 weeks and 12 weeks
  4-item Anxiety short form. Each question is scored ranging from 1 (Never) to 5 (Always). Total raw scores range from 4-20. A lower score indicates low anxiety, a better outcome.
Depression as measured by the PROMIS Depression short form | Baseline, 8 and 12 weeks after enrollment.
  4-item depression short form. Each question is scored ranging from 1 (Never) to 5 (Always). Total raw scores range from 4-20. A lower score indicates low depression, a better outcome.
Mindfulness as measured by the Five Facet Mindfulness Questionnaire | Baseline, 8 and 12 weeks after enrollment.
  15-item mindfulness questionnaire. Each question is scored from 1 (Never or very rarely true) to 5 (Very often or always true). Total raw scores range from 15-75. A higher score indicates more mindfulness, a better outcome.
Physical health as measured by the 6-item Short Form Health Survey within the (SF-12) | Baseline, 8 and 12 weeks after enrollment.
  6 item health survey. The questions vary in scoring and answers with question 1 scores ranging from 1(Excellent) to 5 (Poor). Questions 2-3 scoring ranges from 1 (Yes, limited a lot) to 3 (No, not limited at all). Questions 4-7 scoring ranges from 1 (Yes) to 2 (No). Question 8 scoring ranges from 1 (Not at all) to 5 (Extremely). Questions 9-11 scoring ranges from 1 (All of the time) to 6 (None of the time). Question 12 scoring ranges from 1 (All of the time) to 5 (None of the time).
  Total raw score range from 0-100. A higher score indicates better physical function, a better outcome.
Mental health as measured by the 6-item Short Form Health Survey (SF-12) | Baseline, 8 and 12 weeks after enrollment.
  6 item health survey. The questions vary in scoring and answers with question 1 scores ranging from 1(Excellent) to 5 (Poor). Questions 2-3 scoring ranges from 1 (Yes, limited a lot) to 3 (No, not limited at all). Questions 4-7 scoring ranges from 1 (Yes) to 2 (No). Question 8 scoring ranges from 1 (Not at all) to 5 (Extremely). Questions 9-11 scoring ranges from 1 (All of the time) to 6 (None of the time). Question 12 scoring ranges from 1 (All of the time) to 5 (None of the time).
  Total raw score range from 0-100. A higher score indicates better mental health, a better outcome.
Self-compassion as measured by the Self-Compassion Scale (SCS) | Baseline, 8 and 12 weeks after enrollment.
  26 item compassion scale. Each question is scored ranging from 1 (Almost never) to 5 Almost always). Scoring encompasses subscale measurements of: self kindness (Total raw scores range from 5-25. A high score indicating more self-kindness, a better outcome.), self judgement ( Total raw scores range from 5-25. A low score indicates low self-judgement, a better outcome.), common humanity items (Total raw score range from 4-20. A higher score indicates more common humanity, a better outcome.), isolation (Total raw score range from 4-20. A lower score indicates low feelings of isolation, a better outcome.), mindfulness (Total raw scores range from 4-20. A higher score indicates more mindfulness, a better outcome.), over-identified (Total raw scores range from 4-20. A low score indicates low over-identifying behaviors, a better outcome.)
Educator burnout as measured by the Maslach Burnout Inventory-Educator's Survey | Baseline, 8 and 12 weeks after enrollment.
  22-item Burnout survey for educators. Each question is scored ranging from 0 (Never) to 6 (Every day). Scoring encompasses subcscale measurements of emotional exhaustion (Total raw score range from 0-54. A lower score indicates lower emotional exertion, a better outcome), depersonalization ( Total raw scores range from 0-30. A lower score indicates lower feelings of depersonalization, a better outcome.), and personal accomplishment (Total raw scores range from 0-48 A higher score indicates higher personal accomplishment, a better outcome.)
Acceptability - Satisfaction | Baseline to 8 weeks
  )pen-ended questions regarding barriers and facilitators of adherence and suggestions for improving the MBSR program experience

CONTACTS AND LOCATIONS:
Overall Officials: Martha E Shepherd, DO, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT05051969/ICF_000.pdf